CLINICAL TRIAL: NCT01487655
Title: Waveform Analysis of the Doppler Curve of Ophthalmic Arteries in Primary Open-angle and Normal Tension Glaucoma Patients
Brief Title: Waveform Analysis of the Doppler Curve of Ophthalmic Arteries in Glaucoma Patients
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S271111
Record Dates: First submitted 2011-11-29; First posted 2011-12-07 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2011-09

CONDITIONS: Open-angle Glaucoma; Low Tension Glaucoma
Keywords: Open-angle glaucoma; Low tension glaucoma; Color Doppler Imaging
MeSH Terms: conditions — Glaucoma, Open-Angle; Low Tension Glaucoma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- healthy age matched controls
- normal tension glaucoma patients
- primary open angle glaucoma patients

SUMMARY:
Color Doppler Imaging (CDI) has been providing information about ocular blood flow over the past decades. This non-invasive procedure based on ultrasound technique has identified increased resistance and decreased systolic blood velocities to exist in the ophthalmic arteries of glaucoma patients. However, existing data has provided very little information regarding the analysis of the Doppler waveform in itself and to whether variables such as early systolic acceleration or systolic/diastolic velocity ratios are of any significance in glaucoma disease. In other medical specialties using CDI technology, such as nephrology or cardiology for instance, this analysis has been part of the normal routine. This information has been used in screening patients for disturbed circulation such as arterial stenosis or providing information regarding prognosis of renal and hepatic transplants have been used for decades now.

What is the normal characteristics of the waveform Doppler analysis? To answer this, the investigators will create a normative database using healthy controls.

Are there signs of altered stiffness or compliance in the ophthalmic arteries of glaucoma patients? To answer this, the analysis of early acceleration acceleration and detection of an early peak systolic will be done on the Doppler curves of glaucoma patients and compared to the healthy normative database.

Are there any difference between the two types of glaucoma [primary open-angle glaucoma (POAG) and normal-tension glaucoma (NTG)]? The investigators will compare the variables of the ophthalmic artery waveform in these two groups.

Do any of these Doppler waveform variables have any clinical significance? To answer this, the investigators will search for the existence of any correlation between the waveform data and both functional (visual field testing) and structural (Confocal scanning laser ophthalmoscopy - CSLO) variables of the glaucoma groups.

DETAILED DESCRIPTION:
1. Color Doppler imaging of the ophthalmic artery will be performed 2. Visual field testing will be done 2. CSLO will be done

ELIGIBILITY:
Inclusion Criteria:

* • individuals over 18 years old

  * willing to sign an informed consent and able to comply with the requirements of the study
  * having no other ocular diseases besides glaucoma

Exclusion Criteria:

* • history of ocular trauma

  * intraocular surgery (except for cataract surgery)
  * eye disease (except glaucoma)
  * systemic diseases with ocular involvement like diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Early Systolic Acceleration as a measure of vascular disfunction of the ophthalmic arteries in glaucoma patients | hospital stay, average 3 hours
  Color Doppler Imaging of the ophthalmic artery will provide the waveform of the vessel. There will be a operator-dependent identification of the slope at the beggining of the cardiac cycle and a quantification of the early systolic acceleration. This numberical data will then be compared between healthy and glaucoma groups. Such variables will further be compared to the clinical data (functional - visual field defects and structural - CSLO).

SECONDARY OUTCOMES:
Ratio between systolic and diastolic blood flow velocities as a measure of arterial compliance of the ophthalmic artery in glaucoma patients | Hospital stay, average 3 hours
  Using the CDI-provided ophthalmic artery waveform, there will be an operator-dependent analysis of systolic and diastolic mean blood flow velocities. the ratio between these two variables will be calculated and the numerical data obtained will be compared between the healthy and glaucoma groups. Such ratio will furthermore be compared to functional and structural damage (visual field damage and CSLO, respectively).

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Stalmans, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Department of Ophthalmology, UZLeuven, Leuven, Belgium